CLINICAL TRIAL: NCT04091997
Title: Macrophage Migration Inhibitory Factor for Diagnosing Endometriosis and Its Severity
Status: Completed | Type: Observational
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Sahar MY Elbaradie, associate Professor, Fayoum University Hospital
Other Study IDs: fayoum UH
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Endometriosis
Keywords: Macrophage migration inhibitory factor; Endometriosis; Laparoscopy
MeSH Terms: conditions — Endometriosis | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endometriosis: laparoscopy and directed biopsy of lesions serum macrophage migration inhibitory factor ELIZA assay
  Interventions: Diagnostic Test: serum Eliza assay
- control: diagnostic laparoscopy serum macrophage migration inhibitory factor ELIZA assay
  Interventions: Diagnostic Test: serum Eliza assay

INTERVENTIONS:
Diagnostic Test: serum Eliza assay — laparoscopy and biopsy of lesions in endometriotic patients and seum ELIZA assay of microphage migration inhibitory factor
  Other Names: laparoscopy

SUMMARY:
Endometriosis is a chronic disease affecting women of reproductive age. Macrophage migration inhibitory factor (MIF) is one of non-invasive blood biomarker that was detected in sera of endometriotic patients.The aim of this study was to evaluate the value of serum macrophage migration inhibitory factor in diagnosing endometriosis in women with infertility and chronic pelvic pain and correlate its level with the stage of the disease. Three hundred patient candidate for diagnostic laparoscopy were included in a case-control observational study

DETAILED DESCRIPTION:
observational case-control study conducted in Fayoum University hospital from March 2016 till September 2018. Three hundred women candidate for diagnostic laparoscopy for either infertility or gynecologic chronic pelvic pain were included. The study group included patients with diagnostic criteria of endometriosis. The control group included other causes of infertility or pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* postmenstrual women
* in childbearing period,
* presenting with either gynecologic chronic pelvic pain (CPP) or infertility
* indicated and fit for diagnostic laparoscopy.
* All women must have no hormonal treatment for the last 3 months and.

Exclusion Criteria:

* Women with bleeding tendency,
* suspicious of gynecologic malignancy or
* active infection

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Both groups were comparable regarding the baseline characteristics. these included age, parity, Body mass index, symptoms, type of infertility and chronic pelvic pain
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
level of serum macrophage migration inhibitory factor and stage of the disease | one year
  serum MIF is a promising marker for noninvasive diagnosis of severity of endometriosis

IPD SHARING:
Plan to Share IPD: Undecided